CLINICAL TRIAL: NCT01935375
Title: Multidisciplinary Model of Nurse Midwife Psychotherapy for Postpartum Depression
Brief Title: Multidisciplinary Model of Nurse Midwife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Barbara Posmontier, Assistant Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18981
Record Dates: First submitted 2010-05-24; First posted 2013-09-05 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Postpartum Depression
Keywords: Postpartum Depression; Nurse Midwife; Interpersonal Psychotherapy
MeSH Terms: conditions — Depression, Postpartum | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNM Interpersonal Psychotherapy (Experimental): CNM Interpersonal psychotherapy
  Interventions: Behavioral: CNM Interpersonal Psychotherapy
- Treatment as Usual (Active Comparator): Treatment as Usual is psychotherapy with a mental health provider
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: CNM Interpersonal Psychotherapy — Eight Weekly 50 minute sessions CNM Interpersonal Psychotherapy
  Arms: CNM Interpersonal Psychotherapy
Behavioral: Treatment as Usual — Treatment as Usual is psychotherapy provided by a mental health provider
  Arms: Treatment as Usual

SUMMARY:
HYPOTHESES:

The hypotheses are that:

1. nurse midwives will be able to safely deliver interpersonal psychotherapy by telephone to women with postpartum depression
2. women receiving interpersonal psychotherapy will have less symptoms of postpartum depression, better functioning, better bonding with their babies, and better relationships with their partners
3. women with postpartum depression will be more satisfied with their care than women in the group that was referred to a mental health center.

DETAILED DESCRIPTION:
The specific aims of this pilot non-randomized clinical trial are to evaluate among women with PPD recruited between 6 and 24 weeks postpartum:

1. The (a) feasibility, (b) acceptability and (c) safety of a psychological intervention (Interpersonal Psychotherapy [IPT]) provided by nurse midwives in collaboration with a mental health team (psychiatrist team leader and a licensed social worker) for treatment of PPD in a pilot two-armed non-randomized clinical trial.
2. The preliminary evidence of efficacy of IPT in decreasing depressive symptoms when administered via telephone by nurse-midwives/ women's health nurse practitioner
3. The proposed study will also evaluate preliminary evidence for the efficacy of IPT administered by nurse midwives in

   1. Improving the general level of maternal functioning
   2. Specific improvement in marital adjustment
   3. Increase in maternal infant bonding

This pilot study is the first step in developing an intervention to decrease depressive symptoms, improve functioning, improve interpersonal relationships between mother and spouse and infant, improve access to care, and improve treatment engagement among postpartum women diagnosed with PPD. The intervention will be cost-effective, brief and acceptable to both patients and nurse midwives for incorporation into current midwifery practice. If the IPT program is found to be feasible, acceptable and safe with preliminary evidence of efficacy, a postpartum IPT manual for advanced practice nurses will be finalized in order to test whether other advanced practice nurses such as pediatric nurse practitioners and family nurse practitioners can also safely and effectively administer IPT in a full-scale randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* 6 to 24 weeks postpartum
* 16 years and older
* English-speaking
* Have access to a telephone
* Consents to enter the trial
* Postpartum onset of postpartum depression
* Current use of antidepressant medication as long as dose does not have to be adjusted by subject's healthcare provider during clinical trial

Exclusion Criteria:

* Infant complications requiring medical care beyond 6 weeks postpartum
* Infant birth defects
* Infant being placed for adoption by 6 weeks postpartum
* Maternal mental retardation
* Current use of antidepressant medication that requires dosage adjustment by subject's healthcare provider during clinical trial
* Diagnosis of depression prior to postpartum period
* Active substance or alcohol abuse or dependence
* Active suicidality, homicidality, or current psychosis as assessed by the MINI
* Disabling pain that interferes with the ability to carry out activities of daily living
* Concurrent serious medical co-morbidities (e.g. active lupus, multiple sclerosis, severe cardiac disease severe hypertension, cancer, etc).

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for depression | 12 weeks
  Measure of depression severity

SECONDARY OUTCOMES:
Global Assessment of functioning | 12 weeks
  Measure of functional status
Dyadic Adjustment Scale | 12 weeks
  Measure of dyadic adjustment of marital couple
Social Support Questionnaire | 12 weeks
  Measure of improvement in social support
Client Satisfaction Questionnaire | 12 weeks
  Measure of client satisfaction with midwife counseling
Edinburgh Postnatal Depression Scale | 12 weeks
  Measure of severity of postpartum depression

CONTACTS AND LOCATIONS:
Overall Officials: Barbara E Posmontier, PHD, Principal Investigator — Drexel University; Richard Neugebauer, PhD, Principal Investigator — Columbia University; Scott Stuart, MD, Principal Investigator — University of Iowa; Rita Shaughnessy, PhD, MD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States